CLINICAL TRIAL: NCT03619187
Title: A Phase 3, Open-label, Multicenter Study to Evaluate the Effect of Ivabradine on Exercise Capacity in Heart Transplant Recipients With Elevated Resting Heart Rate
Brief Title: An Interventional Study to Evaluate the Effect of Ivabradine on Exercise Capacity in Heart Transplant Recipients
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20180037
Record Dates: First submitted 2018-08-02; First posted 2018-08-07 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Heart Transplantation, Elevated Resting Heart Rate
MeSH Terms: interventions — Ivabradine

STUDY DESIGN:
Intervention Model Description: This is an open-label, single-arm, multicenter study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Study Product
  Interventions: Drug: Ivabradine

INTERVENTIONS:
Drug: Ivabradine — Ivabradine will be provided in bottles (60 tablets per bottle) labeled ivabradine 5 mg and ivabradine 7.5 mg. The 2.5 mg dose of ivabradine will be achieved by subjects splitting the 5 mg tablets into equal halves.
  Other Names: Corlanor

SUMMARY:
The hypothesis is that the treatment with ivabradine will increase pVO2 after 16 weeks of treatment compared to baseline in the heart transplant recipient population with elevated resting HR.

DETAILED DESCRIPTION:
The primary goal of this study is to assess the impact of ivabradine on cardiopulmonary exercise capacity in heart transplant recipients with elevated resting heart rate (HR).

Exercise capacity will be assessed by the determination of the peak oxygen consumption (pVO2) during standard cardiopulmonary exercise test before and after the treatment period with ivabradine. The secondary goal is to determine HR reduction with ivabradine in the patient population.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent/assent prior to initiation of any study-specific activities/procedures
* Male or female, ≥ 18 to ≤ 70 years of age at signing of informed consent
* History of heart transplantation within 1 to 4 years from screening
* Sinus rhythm and elevated resting HR > 95 bpm at screening (ECG)
* Able to perform exercise testing as required per protocol, per the investigator, at time of screening
* Peak VO2 < 70% of the predicted normal value for age and gender with respiratory exchange ratio (RER) ≥ 1.05, from a CPET conducted during screening

Exclusion Criteria:

* Participation in a cardiac rehabilitation program during the study period
* Treatment for heart transplant rejection within the previous 3 months before screening
* Severe allograft vasculopathy limiting the tolerance of CPET at time of screening
* During CPET at screening, significant adverse finding (eg, exercise-induced early ischemic changes, abnormal blood pressure response, unexpected arrhythmia or other serious finding) that precludes safe participation in the study, per investigator
* Sick sinus syndrome, sinoatrial block and/or third degree atrioventricular block, unless a functioning demand pacemaker is present, or pacemaker dependency at screening
* Resting systolic blood pressure >160 mmHg or <100 mmHg, or diastolic blood pressure >90 mmHg at screening
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion
* Presence of clinically meaningful acute or chronic infection, per investigator, at screening
* Major medical event or procedure (as determined by investigator) within 3 months prior to screening
* Previously received ivabradine after heart transplantation (prior to the participation in this study)
* Subjects taking QT prolonging medicinal products for cardiovascular (eg, but not limited to, quinidine, disopyramide, bepridil, sotalol, ibutilide) or non-cardiovascular disease (eg, but not limited to, pimozide, ziprasidone, sertindole, mefloquine, halofantrine, pentamidine, cisapride, intravenous (IV) erythromycin)
* Subjects should not be receiving beta-blockers, diltiazem, or verapamil for at least 7 days before screening
* Subjects exposed to a strong Cytochrome P450 3A4 (CYP3A4) inhibitor (examples of strong CYP3A4 inhibitors include; azole antifungals [eg, itraconazole], macrolide antibiotics [eg, clarithromycin, telithromycin], human immunodeficiency virus protease inhibitors, [eg, nelfinavir], and nefazodone]) within 14 days prior to screening, or to a strong CYP3A4 inducer (examples of CYP3A4 inducers include; St. John's wort, rifampicin, barbiturates, and phenytoin) within 28 days prior to screening
* Currently receiving treatment in another investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded.
* Hemoglobin < 8 g/dL at screening (or within 3 months prior to screening if no clinically meaningful event, as determined by the investigator, has occurred in that period) and not expected to receive blood transfusion during the study
* Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2 (by the Modification of Diet in Renal Disease [MDRD] equation) at screening (or within 3 months prior to screening)
* Subject has known sensitivity to any of the products to be administered during dosing
* Female subject is pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 2 weeks after the last dose of investigational product
* Female subjects of childbearing potential unwilling to use 1 highly effective method of contraception during treatment and for an additional 2 weeks after the last dose of investigational product. Refer to Section 12.5 for additional contraceptive information
* Female subjects of childbearing potential with a positive pregnancy test assessed at screening by a serum pregnancy test

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-02 (Estimated); Primary Completion 2020-02-19 (Estimated); Study Completion 2020-02-19 (Estimated)

PRIMARY OUTCOMES:
pVO2 | Week 16
  To evaluate the effect of treatment with ivabradine on exercise capacity as measured by peak oxygen consumption (pVO2)

SECONDARY OUTCOMES:
Resting Heart Rate | Week 16
  To evaluate the effect of treatment with ivabradine on resting heart rate (HR)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com